CLINICAL TRIAL: NCT04442997
Title: Use of Cesarean Birth at Private Health Facilities in Lilongwe and Blantyre, Malawi
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0468; NICHD/K12 HD001271-21 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Cesarean birth

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the research study is to collect preliminary data to which future outcomes after implementing quality improvement projects or research will be compared. There will be observation of the labor and delivery services received and resulting outcomes of women and infants who deliver at private health facilities in urban Malawi. Data will be collected at admission, delivery, and discharge from women and providers on patient characteristics, labor and obstetric characteristics, delivery factors, and pregnancy outcomes that result during the course of the hospitalization. This will include the vital status of the mother and the infant. The overall hypothesis is that cesarean birth rates will be higher than the ecologically supported 10% cesarean birth rate, and that there may be cesareans that are performed without clear medical indication.

DETAILED DESCRIPTION:
Background:

Cesarean birth is the most commonly performed surgery in the world. It is a major abdominal procedure that can save maternal and perinatal lives when properly indicated, but when performed without medical necessity, is associated with adverse outcomes. Global cesarean birth rates are increasing, but there has been a less pronounced rise in sub-Saharan Africa (SSA) where rates tend to be below 5.0%. However, in Sub-Saharan Africa (SSA) and other low- and middle-income countries (LMIC), there is a recognition that significant in-country disparities in the use of cesarean birth exist. Rates are higher in urban settings, and there is evidence that they are higher in private versus public facilities.

Objective and Aims:

The main objective of this prospective, cross-sectional, observational study is to observe the use of cesarean birth at three private health facilities in urban Malawi by the end of the study. This will be achieved by getting an understanding of the current delivery practices and patient characteristics, as well as associated outcomes of women who choose to deliver at these private facilities in order to understand how and under what circumstances the surgery is being used.

Aim 1: Observe prevalence of and indications for cesarean birth in three private health facilities in urban Malawi in the overall cohort and in ten mutually exclusive subgroups defined by the WHO-endorsed Robson Classification for cesarean birth

Aim 2: Determine risk factors associated with cesarean birth among Robson subpopulations of women at study sites, and the distribution of adverse pregnancy outcomes across those subgroups

Aim 3: Identify target modifiable risk factors or areas for potential quality improvement or prospective research studies to optimize the use of cesarean birth within these facilities that may have generalizable implications

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Admitted for delivery or observation

Exclusion Criteria:

-

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women admitted for observation or delivery at 3 private health facilities in Malawi.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of participants using cesarean section delivery as assessed by survey questionnaires | Hospital admission to discharge, about 3-4 days
Types of indications for cesarean birth | Hospital admission to discharge, about 3-4 days

SECONDARY OUTCOMES:
Types of adverse pregnancy outcomes among participants using cesarean section | Hospital admission to discharge, up to 1 week
  The types of adverse pregnancy outcomes reported among participants with cesarean section deliveries will be assessed via survey questionnaires. Data will be reported by population subgroup. Population subgroups will be defined by the World Health Organization-endorsed Robson Classification for Cesarean Birth
Types of risk factors for Cesarean birth | Hospital admission to discharge, about 3-4 days
  The types of modifiable risk factors for cesarean birth reported among participants that use cesarean section delivery will be assessed via survey questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Margo Harrison, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (3):
- Malawi (3):
  - Mwaiwathu Private Hospital, Blantyre
  - Area 18 Medi Clinic - Asamala Health Services, Lilongwe
  - Good Hope Private Clinic, Lilongwe

IPD SHARING:
Plan to Share IPD: No